CLINICAL TRIAL: NCT05921799
Title: A Novel Point-to-care Method for Fast Evaluation of Viscoelastic Hemostasis Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0951
Record Dates: First submitted 2023-06-18; First posted 2023-06-27 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2023-06

CONDITIONS: Perioperative Period
Keywords: blood coagulation; blood coagulation tests
MeSH Terms: conditions — Thrombosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General anesthesia Patients: Subjects experiencing general anesthesia such that viscoelastic testing is performed to assess coagulopathy.
  Interventions: Procedure: Blood specimen collection

INTERVENTIONS:
Procedure: Blood specimen collection — Routinely collect citrate blood and native blood from patients as required by their condition.

SUMMARY:
This study compares the results of the existing coagulation monitoring technology to the Ultrasound-based viscoelastic hemostasis analysis, a new method, using small amount of extra blood obtained during routine blood draws in surgery patients.

DETAILED DESCRIPTION:
Ultrasound-based viscoelastic hemostasis analysis is a novel POC diagnostic method, which is suitable for use in surgical care settings.

The novel viscoelastic hemostasis analysis uses ultrasound guided waves to characterize the dynamic changes in viscoelastic properties of a blood sample during coagulation and clot lysis, which will be the surgical assay for monitoring hemostasis during major surgical procedures in adult patients.

This single-center, prospective, observational pilot study will evaluate the analytical performance as well as compared to standard coagulation tests and comparable measures using conventional viscoelastic testing methods.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled for surgery with general surgery
* Subject is 18 years or order
* Subject requires routine TEG measurement

Exclusion Criteria:

* Subject is unwilling to participate
* Subject is unable to sign a consent form
* Subject is unsuitable for blood drawing
* Subject is unsuitable for this study in the opinion of the anesthesiologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants for this study will be recruited at the Second Affiliated Hospital Zhejiang University School of Medicine. The study participants will be adult general anesthesia patients such that viscoelastic testing is performed to assess coagulopathy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of the novel viscoelastic hemostasis analysis results to TEG results | 1 day
  Coagulation function assessed by the novel viscoelastic hemostasis analysis and TEG
Comparison of the novel viscoelastic hemostasis analysis results to standard coagulation test results | 1 day
  Coagulation function assessed by the novel viscoelastic hemostasis analysis and standard coagulation test

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University anesthesiology department, Hangzhou, Zhejiang, China